CLINICAL TRIAL: NCT02932163
Title: Relationships Between Muscular Impairments, Pain, and Disability in Patients With Chronic Non-specific Low Back Pain: a Cross Sectional Study
Brief Title: Predictors of Chronic Non-specific Low Back Pain
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: chronic non-specific LBP
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; disability; endurance
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic non-specific low back pain (CNSLBP) has been defined as a persistent pain in the lower back for at least three months with no known causes. The CNSLBP prevalence is estimated of 90% among all types of the LBP. The LBP imposes high direct and indirect costs on the patients and the society. Whereas a specific pathology has not been identified for CNSLBP, mechanical factors (e.g. changes in muscle length, strength, or endurance) may contribute to the pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic non-specific LBP,
* LBP duration ≥ 6 months.

Exclusion Criteria:

* spinal osteoarthritis,
* spondylolisthesis,
* history of vertebral fractures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non-specific LBP were recruited from five hospitals in Ahvaz, Iran.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change of Pain intensity | Baseline
  Visual Analogue Scale
Change of Disability | Baseline
  Oswestry disability index

CONTACTS AND LOCATIONS:
Overall Officials: JORGE H VILLAFAÑE, PhD, Principal Investigator — IRCCS Don Gnocchi Foundation

IPD SHARING:
Plan to Share IPD: No